CLINICAL TRIAL: NCT06138457
Title: The ECOSTRESS Study: Influence of the Objective Structured Clinical Examination on Stress Among Medical Student
Acronym: ECOSTRESS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2023BOUILLON-MINOIS-ECOSTRESS
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Heart Rate Variability; Stress; Medical Student
Keywords: stress; exam; medical student; heart rate variability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will assess stress using heart rate variability during examination on medical student. Three time of measurement will be performed. First standardized objective clinical examination, second classic table examination and third a control day.

DETAILED DESCRIPTION:
French medical students have benefited from a new evaluation method since 2020 in the form of a standardized objective clinical examination (OSCE). This examination consists of an evaluation of an initial clinical situation, in relation to a pre-identified and nationally identical objective in all Medical School. During these exams, the student has one minute of preparation then seven minutes of evaluation in front of a facilitator, member of the teaching staff. An examiner is also present in the room to search in real time for keywords intended for grading. The examiner and facilitator may or may not be tenured teachers. Students benefit from annual training organized by the Medical School of Clermont-Ferrand in which they all participate. This exam appears to be excessively stressful for students. However, there is currently no data regarding the objective measurement of the stress of these students. Heart rate variability is a biomarker of stress measured with a simple heart rate monitor or a watch, completely painless, non-intrusive, and used by the general public routinely in many areas (monitoring sports sessions, etc...).

ELIGIBILITY:
Inclusion Criteria:

* All medical student that agree to participate

Exclusion Criteria:

* All medical student that disagree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical student between fourth and sixth year of med school
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2030-06-29 (Estimated); Study Completion 2030-06-29 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | 24 hours
  Comparison of heart rate variability during one day of OSCE versus a traditional table examination.

SECONDARY OUTCOMES:
Sociodemographic | Once
  Study of factors influencing heart rate variability (time of passage, anticipatory stress, sociodemographic, or lifestyle habits).
Subjective stress | 12 hours
  Study of stress using visual analogic scale (VAS)
Stress correlation | Once
  Study of correlation between subjective stress (VAS) and objective stress (HRV)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste BOUILLON-MINOIS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Medical School of Clermont-Ferrand, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - CHU clermont-ferrand, Clermont-Ferrand